CLINICAL TRIAL: NCT06467136
Title: Motor Imagery for Treatment Enhancement and Efficacy (MI-TEE) in Persons With Apraxia of Speech
Brief Title: Motor Imagery for Treatment Enhancement and Efficacy in Persons With Apraxia of Speech
Acronym: MI-TEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Lauren Bislick Wilson, Associate Professor; Director UCF Aphasia House, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AWD00005714; 1R21DC020548-01A1 (NIH)
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-06

CONDITIONS: Apraxia, Oral; Apraxia of Speech
Keywords: Treatment of Apraxia of Speech; Home Practice for Apraxia of Speech; AOS; Apraxia of speech
MeSH Terms: conditions — Apraxias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A research assistant will be blind to study condition and time point
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Condition 1 (Experimental): Condition 1 will have three phases: (A) no treatment; (B) speech therapy alone; (C) speech therapy plus MI-TEE (the home practice program).
  Interventions: Behavioral: Sound production treatment; Behavioral: Motor Imagery Practice
- Condition 2 (Experimental): Condition 2 will include two phases: (A) no treatment; (C) speech therapy plus MI-TEE (the home practice program).
  Interventions: Behavioral: Sound production treatment; Behavioral: Motor Imagery Practice

INTERVENTIONS:
Behavioral: Sound production treatment — Evidence based treatment for apraxia of speech, developed by Julie Wambaugh.
  Other Names: SPT
Behavioral: Motor Imagery Practice — Practice of target items using motor imagery during home practice

SUMMARY:
Treatment of post-stroke apraxia of speech (AOS) requires frequent and ongoing practice with a speech-language pathologist to facilitate lasting behavioral change, which is costly and, therefore, inaccessible to many patients. Thus, there is a critical need to identify novel, cost-effective ways to supplement speech therapy to increase opportunities for practice and optimize treatment outcomes. Our long-term goal is to develop an effective, home-practice, computer-based, motor imagery protocol Motor Imagery for Treatment Enhancement and Efficacy (MI-TEE) which will serve as an adjunct to routine speech therapy to optimize treatment response in persons with AOS. The overall objectives of this application are to (i) evaluate the acceptability and feasibility of MI-TEE as a home practice program and (ii) determine the efficacy of MI-TEE with speech therapy, compared to speech therapy alone, in improving speech production in people with AOS. Our central hypothesis is that MI-TEE will be an accessible, feasible, and efficacious adjunct to speech therapy. To attain our objectives, the following specific aims will be pursued using two single-subject experimental designs with multiple baselines across participants (n=18): 1) Evaluate the acceptability and feasibility of MI-TEE as an adjunct to speech therapy for the rehabilitation of AOS; and 2) Compare the efficacy of adjunctive MI-TEE plus standard speech therapy to standard speech therapy alone. Under the first aim, observational data, surveys, and semi-structured interviews will be employed to assess the acceptability (perceived satisfaction, appropriateness, and intent to continue use) and feasibility (recruitment, retention, and intervention adherence rates) of MI-TEE. For the second aim, accuracy of articulation for trained words and untrained words (generalization) will be measured pre-treatment, repeatedly during the treatment phase, and post-treatment. Improvements in speech accuracy will be documented using a binary scoring system (correct/incorrect). Multilevel analyses will be used to address rate of acquisition, overall change, and response variation across participants.

DETAILED DESCRIPTION:
This R21 Proposal will employ a mixed-methods design in 18 individuals with apraxia of speech and mild-moderate co-occurring aphasia to examine two Aims:

Aim 1. Evaluate the acceptability and feasibility of MI-TEE as an adjunct to speech therapy for the rehabilitation of AOS. This Aim will Incorporate observational data, survey responses (self-report) and semi-structured interviews. Specifically, mixed quantitative and qualitative methods will be employed to assess the acceptability and feasibility of MI-TEE. Quantitative data will include observational data and results of survey responses. Qualitative data will include themes that emerge from open-ended survey items and semi-structured interviews. Assessment of acceptability will occur after completion of the 12-week treatment program. Participants will meet individually with a member of the research team to complete acceptability surveys and semi-structured interviews. Acceptability data will include perceived satisfaction, perceived appropriateness, and intent to continue use. Assessment of feasibility will determine the extent to which the treatment, including study design and procedures, is executed effectively. Feasibility data will be collected by research staff and will include recruitment feasibility (percent of eligible individuals agreeing to participate), retention rate, and adherence rates (ability of participants to adhere to MI-TEE).

Aim 2. Compare the efficacy of adjunctive MI-TEE to standard speech therapy (Sound Production Treatment) alone. This aim will employ a single subject experimental design (SSED) with multiple baselines across participants and probes across behaviors will be used to explore the effects of speech therapy alone compared to speech therapy with MI-TEE in 15 stroke survivors with AOS. The treatment design will include multiple phases: (A) no treatment; (B) speech therapy alone; (C) speech therapy plus MI-TEE. The first "A" will consist of pre-treatment baseline testing, while the second will consist of maintenance testing. Following baseline probes, treatment probes will be extended sequentially to each of the two lists of stimuli, which are described in the following section (Experimental Stimuli). Probing will continue throughout the treatment phases. After cessation of all treatment, follow-up probes will be conducted at 2, 6, and 10 weeks. Accuracy of articulation of two lists of experimental stimuli will be measured repeatedly via probes.

This proposal will include 18 adult (≥18 years of age) stroke patients. No subpopulation of adults with apraxia of speech and aphasia will be excluded (see Inclusion of Women and Minorities).

Potential participants will have had a left hemisphere stroke (documented by imaging with either CT or MRI) and be 6 months or more post-stroke, right handed, English as a primary language, high-school education or equivalent, between the ages of 18 and 90, pass a hearing screening at 35 dB hearing level (HL) at 500, 1K, and 2K Hz for at least one ear, and have normal or corrected to normal visual acuity as determined by a vision screen (Tumbling E eye chart).

Participants must demonstrate AOS. To elicit speech samples from which to judge presence/absence of AOS characteristics subtests I, II, IV, and V of the Apraxia Battery for Adults - second edition (ABA- 2) will be administered, along with word and sentence repetition tasks and a diagnosis of AOS will be based on the presence of primary clinical characteristics including 1) slow speech rate characterized by lengthened segment and intersegment durations, 2) sound distortions, 3) distorted sound substitutions, and 4) prosodic abnormalities. Two experienced speech-language pathologists (SLPs) must agree upon the presence of AOS. Co-occurring aphasia will be determined by the presence of multimodal language processing deficits, as measured by the Comprehensive Aphasia Test. Individuals with aphasia must demonstrate sufficient auditory comprehension (i.e., follow one-step commands or greater) to participate in treatment.

Severity of AOS will be assessed by two experienced SLPs via consensus ratings. SLPs will watch audiovisual recordings of participants completing subtests from the ABA-2. Included participants must demonstrate a minimum ability to produce single sounds, but must not be too mild that sound errors occur infrequently. In addition, the Apraxia of Speech Rating Scale as a clinical composite measure of perceived speech severity.

Procedures. Participants, once recruited, will be interviewed as part of an (IRB-approved) intake and informed consent process. During this initial meeting, a member of the research team will gather preliminary personal identifying information (PII) and study-related neurological health information (see item Ia above). Additionally, medical records will be requested after an IRB-approved HIPAA-authorization/release of records has been obtained from participants to confirm neurologic diagnosis.

Participants' PII will be protected by the assignment of an alpha-numeric code to study data files, and all paper PII (intake and informed consent forms) will be locked in a file drawer to be accessed only by the PI and authorized lab personnel. Additionally, digital PII files will be password protected, with a password known only to the PI and authorized lab personnel. All PII will be destroyed one year following the completion of the research study.

Following intake and informed consent process, participants will undergo stimulability testing to determine treatment targets. Specifically, participants will be asked to repeat several words of varying lengths and difficulty. Participant responses will be audiovisually recorded and analyzed offline by student researchers, under the supervision of the PI, to identify treatment targets. Once treatment targets have been identified the research team can create treatment stimuli and probes. Prior to the initiation of treatment participants will undergo baseline testing. A minimum of five baseline data points will be collected prior to the initiation of treatment. Repeated probes will be administered after every two hours of therapy, immediately following treatment termination and at follow-up (2-, 6-, and 10-weeks post treatment). Participant performance on the probe data will be audiovisually recorded for scoring by blinded members of the research team. All audiovisual recordings of participant responses will be saved and filed using the assigned alpha-numeric code.

All study participants will receive speech therapy 3 days a week for 8.3 weeks for 50 minutes a day. Speech therapy will take place at the UCF Innovation Center and/or in the participants' home if they are unable to commute to UCF. Speech therapy will consist of Sound Production Treatment (SPT), an established and evidence-based treatment for post-stroke AOS.

MI-TEE is a computer-based, home-practice protocol that provides additional opportunities to practice words targeted during speech therapy. Participants will be instructed to complete the MI-TEE protocol 3 times a week, on non-treatment days, for 20-30 minutes to practice words and sounds addressed in speech therapy. Participants will use MI-TEE to practice lists of 24 target words (i.e., the trained lists). During the MI-TEE practice sessions, participants will be instructed to sit at a desk with a computer or tablet, equipped with a webcam, in a quiet room in their home, with a power outlet, and without distractions. An audiovisual recording of a person's mouth producing a word trained during the SPT session (treatment stimuli) will play one time on the screen. Following the presentation of the stimuli, participants will be asked to "imagine speaking the whole word" in their mind without moving any articulators or producing any sounds. They will be told that they should feel the movement of the specific articulators associated with the physical pronunciation of each sound in the word. A two-week training period will be provided, during which study staff will give live feedback via Zoom while patients engage in MI-TEE from their home. After the training period, MI-TEE sessions will be recorded and viewed offline by research staff to assess adherence. Research staff will visit participants in their homes prior to the start of the study to assist with equipment set-up and will check in virtually (or in person if physical changes are required) periodically over the course of the study to address any technical needs. If needed the following materials will be provided to the participant for the duration of the study: computer (laptop) or tablet, webcam, a power extension cord, noise cancelling headphones.

Assessment of acceptability will occur after completion of the 8.3-week treatment program. Participants will meet individually with a member of the research team to complete acceptability surveys and semi-structured interviews. Acceptability data will include perceived satisfaction, perceived appropriateness, and intent to continue use. Caregivers will also be invited to participate in the surveys and semi-structured interviews. Assessment of feasibility will determine the extent to which the treatment, including study design and procedures, is executed effectively. Feasibility data will be collected by research staff and will include recruitment feasibility (percent of eligible individuals agreeing to participate), retention rate, and adherence rates (ability of participants to adhere to MI-TEE). To assess participant adherence to the protocol, all MI-TEE sessions will be recorded for review by research staff offline and a procedural checklist will be used to calculate treatment fidelity. Feedback will be provided on a weekly basis if deviation from the protocol is observed. Feasibility data will be collected by research staff throughout the study.

Planned Analysis Quantitative data will be summarized using descriptive statistics (frequencies, percent, mean, standard deviation, range). Semi-structured interviews will be transcribed for content and will undergo domain and taxonomic analyses to identify themes reflecting participant perspectives on the accessibility, feasibility, and use of MI-TEE, and their overall experience. Domain analysis will also be employed for open-ended survey responses. The two sources of qualitative data will be triangulated with the statistical analyses of quantitative data to determine feasibility and acceptability aspects of recruitment, data collection, and intervention procedures.

Assessment of treatment effects will match that of previous investigations by Bislick and Wambaugh and will include effect size measures and AOS benchmarks. Additionally, multilevel analyses will be performed to address rate of acquisition, overall change, and response variation across participants. Successful adoption of multilevel models has increased in single case designs, and they have shown to be quite powerful with samples as small as three cases. The number of participants requested in this study is larger than most of the published investigations on SPT, including those that have compared different treatment protocols via SSED, and is sufficient for this preliminary investigation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 90 yrs. old
* At least 6 months post left hemisphere stroke
* Demonstrate AOS
* Speak English as their primary language
* Pass a hearing screening at 35 dB HL at 500, 1K, and 2K Hz for at least one ear
* Normal or corrected to normal visual acuity

Exclusion Criteria:

* Unable to follow two-step commands and greater than moderate aphasia
* Moderate - severe dysarthria
* Untreated depression or other psychiatric illness
* Degenerative neurological illnesses
* Less than 3 on the MIQ-RS77
* Less than a 4 on 3/5 domains on the FACETS
* Less than a 23 on the Raven's Coloured Progressive Matrices
* Receive other speech therapy while participating in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Assessment of acceptability will occur after completion of the 8.3 week treatment program
  Participants will complete acceptability surveys and meet individually with a member of the research team to engage in semi-structured interviews.82 Acceptability data will include perceived satisfaction and appropriateness, experience with MI-TEE, and intent to continue use.
Recruitment feasibility | Through study completion, up to 24 weeks.
  Feasibility data will be collected by research staff throughout the study and will include recruitment feasibility, the percent of eligible individuals agreeing to participate in the MI-TEE program.
Adherence rates | Start of MI-TEE program to the end of the 8.3 week treatment program for each participant.
  Feasibility data will be collected by research staff throughout the study and will include adherence rates, the participants ability to adhere to the MI-TEE protocol.
Retention rate | Start of MI-TEE enrollment to the end of the 8.3 week treatment program for each participant.
  Feasibility data will be collected by research staff throughout the study and will include retention rates, the percent of participants who complete the entire MI-TEE program.
Rate of change | From enrollment to the end of maintenance at 10 weeks, total of up to 23 weeks.
  The dependent variable is rate of change for accuracy of sound production in experimental words produced during probes.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Bislick Wilson, Ph.D., Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida Innovation Rehabilitation Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share de-identified participant outcomes via publication and conference presentations.
Supporting Information: Study Protocol, SAP
Time Frame: After study completion. Available via supplemental materials in publications.
Access Criteria: Access to peer-reviewed/published manuscripts